CLINICAL TRIAL: NCT01394666
Title: Treatment Patterns and Associated Outcomes in Chronic Phase (CP) Chronic Myelogenous Leukemia (CML) Patients Who Fail Imatinib 400 mg Daily
Brief Title: Non-interventional Treatment Patterns Study in Chronic Phase Chronic Myelogenous Leukemia (CP-CML)
Status: Completed | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: CA180-240
Record Dates: First submitted 2011-07-08; First posted 2011-07-14 (Estimated); Last update posted 2016-07-11 (Estimated); Status verified 2016-07

CONDITIONS: Chronic Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- CP-CML patients who have failed Imatinib 400 mg daily

SUMMARY:
The purpose of this study is to evaluate treatment patterns and associated outcomes for CP-CML patients who fail Imatinib 400 mg daily in a real-world setting.

DETAILED DESCRIPTION:
Time Perspective: Retrospective and Prospective

ELIGIBILITY:
For more information regarding BMS clinical trial participation, please visit www.BMSStudyConnect.com.

Inclusion Criteria:

* Adult patients (18 years or older) in Chronic phase CML patients who have been treated with Imatinib 400 mg and have failed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary care clinic, academic and community oncology centers
Sampling Method: Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2011-05; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Complete Cytogenic Response (CCyR) for CP-CML patients who failed Imatinib 400 mg daily | At 3 months post treatment change
Complete Cytogenic Response (CCyR) for CP-CML patients who failed Imatinib 400 mg daily | At 6 months post treatment change
Complete Cytogenic Response (CCyR) for CP-CML patients who failed Imatinib 400 mg daily | At 12 months post treatment change

SECONDARY OUTCOMES:
Prognostic factors (clinical and demographic characteristics) that influence treatment selection for CP-CML patients who fail imatinib 400 mg daily | Baseline
Prognostic factors (clinical and demographic characteristics) that influence treatment selection for CP-CML patients who fail imatinib 400 mg daily | 3 months after start of treatment
Prognostic factors (clinical and demographic characteristics) that influence treatment selection for CP-CML patients who fail imatinib 400 mg daily | 6 months after start of treatment
Prognostic factors (clinical and demographic characteristics) that influence treatment selection for CP-CML patients who fail imatinib 400 mg daily | 12 months after start of treatment
Best response rates achieved by patients if no CCyR | Baseline
Best response rates achieved by patients if no CCyR | 3 months after start of treatment
Best response rates achieved by patients if no CCyR | 6 months after start of treatment
Best response rates achieved by patients if no CCyR | 12 months after start of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb

REFERENCES:
- See also: BMS Clinical Trials Disclosure — http://www.bms.com/clinical_trials/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx
- See also: For FDA Safety Alerts and Recalls refer to the following link: http://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm — http://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm